CLINICAL TRIAL: NCT01969331
Title: An Interventional, Prospective, Multi-center, Double-blind, Placebo Controlled Postmarketing Study to Evaluate Efficacy and Safety of Normia® Probiotic Treatment as a Supportive Therapy in Eradication of H. Pylori
Brief Title: Efficacy and Safety of Probiotic Treatment as a Supportive Therapy in Eradication of H. Pylori
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Goran Hauser (Other)
Collaborators: Jadran Galenski laboratorij d.d.Rijeka (Unknown)
Responsible Party: Sponsor-Investigator, Goran Hauser, Goran Hauser MD, PhD, University Hospital Rijeka
Organization: University Hospital Rijeka (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JGL/02/09
Record Dates: First submitted 2013-10-09; First posted 2013-10-25 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Helicobacter Pylori Infection
Keywords: Gastritis; Helicobacter pylori
MeSH Terms: conditions — Gastritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): maltodextrin, microcrystalline cellulose; hypromellose, silicium dioxide (E551), magnesium stearate, colouring agent: titanium dioxide ( E171) Placebo as an addition to standard H. Pylori eradication therapy 7 days of initial therapy (2 antibiotics + PPI), followed by 21 days of PPI only therapy.
  Two weeks after the end of PPI therapy subjects are seen at the follow up visit.
  Interventions: Dietary Supplement: Placebo
- Normia (Active Comparator): Lactobacillus rhamnosus GG, LGG® and Bifidobacterium, BB-12® Normia® probiotic as an addition to standard H. Pylori eradication therapy 7 days of initial therapy (2 antibiotics + PPI), followed by 21 days of PPI only therapy. One capsule twice per day/14 days Two weeks after the end of PPI therapy subjects are seen at the follow up visit.
  Interventions: Dietary Supplement: Normia

INTERVENTIONS:
Dietary Supplement: Normia — One capsule twice a day/14 days
  Other Names: Lactobacillus rhamnosus GG, LGG® and Bifidobacterium, BB-12®
  Arms: Normia
Dietary Supplement: Placebo — maltodextrin, microcrystalline cellulose; hypromellose, silicium dioxide (E551), magnesium stearate, colouring agent: titanium dioxide ( E171)
  Arms: Placebo

SUMMARY:
The aim of the study is to establish efficacy and safety of Normia® probiotic, used as an add-on therapy in treatment of H. Pylori infection with the standard triple therapy approach.

The primary objective in the study is determination of efficacy of Normia® probiotic as a supportive therapy in achieving a higher percentage of eradication of H. Pylori.

The secondary objectives are to assess:

* Safety profile of Normia® probiotic in everyday use, e.g. reduction in number of side-effects and better compliance to the eradication therapy
* Safety and efficacy of Normia® probiotic in different demographic subgroups

DETAILED DESCRIPTION:
Gastroenterologists and general practitioners have increasingly more possibilities of prescribing probiotic preparations as the only or (more often) adjuvant therapy in certain indications. A significant step forward was made in the current report of the European Helicobacter Study Group ,which states that "Certain probiotics and prebiotics show promising results as an adjuvant treatment in reducing side effects". At this stage,probiotics are classified as Grade D recommendation. That is precisely why the investigators believe that clinical studies are necessary in order for such effects to be objectively proven in a clinical setting.

The investigators decided to conduct a clinical trial based on a clearly defined and sufficiently frequent indication,with a preparation of known probiotic composition that is easily available on the market, and in a real setting where such approach is bound to show both advantages and disadvantages.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed H. Pylori infection.
* Otherwise healthy subjects taking H. pylori eradication therapy.
* Age above 16 years.
* Male and female subjects.
* Subject who provided written informed consent prior to undergoing any study procedure.

Exclusion Criteria:

* Pregnancy or lactation.
* Severe diseases such as malignant diseases, severe renal/liver impairment, HIV infection etc.
* Chronic diseases such as diabetes mellitus, hypertension, epilepsy or atherosclerosis which are under treatment and well regulated are not an exclusion criterion.
* Subject who is not mentally capable of adhering to the protocol.
* Drug addiction or alcoholism.
* Any other clinical condition which, in the opinion of the attending physician, would not allow safe administration of the study medications.
* Subjects participating in any other clinical trial.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 804 (Actual)
Dates: Start 2008-12; Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Percentage of eradication of H.Pylori infection with Normia® probiotic as a additional therapy to standard triple therapy regimen | 40-44 days
  Duration of participation in the study will depend on the duration of therapy prescribed by the attending physician. The exact type of the basic (triple) therapy prescribed to each subject is at the discretion of the physician.
  Assuming standard therapy regimes for this indication, the shortest possible participation in the study will be as follows:
  * 7 days of initial triple therapy, followed by
  * 21 days of PPI therapy only, followed by
  * 14 days +/- 2 days to the follow up visit. Therefore, study participation will take between 40 and 44 days.

SECONDARY OUTCOMES:
Reducing the number of adverse events for H. pylori eradication triple therapy using Normia® probiotic as a supportive therapy | 40-44 days
  Subjects will receive therapy considered to be a "golden standard" for this indication (triple therapy eradication protocol). Subjects receiving Placebo will be receiving standard triple therapy as well.

CONTACTS AND LOCATIONS:
Overall Officials: Goran Hauser, MD,PhD, Principal Investigator — UH Rijeka
Locations (1):
- University Hospital Rijeka, Rijeka, Rijeka, Croatia